CLINICAL TRIAL: NCT02275533
Title: Randomized Phase II Study to Assess the Role of Nivolumab as Single Agent to Eliminate Minimal Residual Disease and Maintain Remission in Acute Myelogenous Leukemia (AML) Patients After Chemotherapy (REMAIN TRIAL)
Brief Title: Testing Nivolumab to Prevent Disease From Coming Back After Treatment in Patients With Acute Myeloid Leukemia, REMAIN Trial
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-02167; NCI-2014-02167 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CIRB 15-0185; CVCIRB 15-0185; 9706 (Other: University of Chicago Comprehensive Cancer Center EDDOP); 9706 (Other: CTEP); N01CM00071 (NIH); P30CA014599 (NIH); UM1CA186644 (NIH); UM1CA186686 (NIH); UM1CA186689 (NIH); UM1CA186691 (NIH); UM1CA186712 (NIH); UM1CA186717 (NIH); ZIABC011078 (NIH)
Record Dates: First submitted 2014-10-24; First posted 2014-10-27 (Estimated); Results first posted 2025-11-06 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Specimen Handling; Biopsy; Watchful Waiting; Observation; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (nivolumab) (Experimental): Patients receive nivolumab IV over 60 minutes once every 2 weeks. Treatment repeats every 2 weeks for 46 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy at screening, months 3, 6, and 12, as clinically indicated, and during off-study evaluation. Patients also undergo collection of blood samples at screening, weeks 9, 13, 25, and 53, and during off-study evaluation or at time of clinically suspected relapse. Patients may undergo ECHO as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Procedure: Echocardiography Test; Biological: Nivolumab
- Arm II (observation) (Active Comparator): Patients undergo standard of care clinical observation for up to 2 years. Upon disease relapse, patients may cross-over to Arm I. Patients also undergo bone marrow biopsy at screening, months 3, 6, and 12, as clinically indicated, and during off-study evaluation. Patients also undergo collection of blood samples at screening, weeks 9, 13, 25, and 53, and during off-study evaluation or at time of clinically suspected relapse. Patients may undergo ECHO as clinically indicated.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Marrow Biopsy; Other: Clinical Observation; Procedure: Echocardiography Test

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Marrow Biopsy — Undergo bone marrow biopsy
  Other Names: Biopsy of Bone Marrow; Biopsy, Bone Marrow
Other: Clinical Observation — Undergo standard of care clinical observation
  Other Names: observation
  Arms: Arm II (observation)
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Biological: Nivolumab — Given IV
  Other Names: ABP 206; BCD-263; BMS 936558; BMS-936558; BMS936558; CMAB819; MDX 1106; MDX-1106; MDX1106; NIVO; Nivolumab Biosimilar ABP 206; Nivolumab Biosimilar BCD-263; Nivolumab Biosimilar CMAB819; ONO 4538; ONO-4538; ONO4538; Opdivo
  Arms: Arm I (nivolumab)

SUMMARY:
This phase II trial studies how well nivolumab works in eliminating any remaining cancer cells and preventing cancer from returning in patients with acute myeloid leukemia that had a decrease in or disappearance of signs and symptoms of cancer after receiving chemotherapy. Immunotherapy with monoclonal antibodies, such as nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate and compare the progression free survival rate after randomization in the two treatment arms (nivolumab versus [vs.] observation).

SECONDARY OBJECTIVES:

I. To determine and compare the overall survival rates in the two arms. II. To determine and compare the incidence of non-relapse mortality in the two arms.

III. To evaluate the toxicities of nivolumab as maintenance.

EXPLORATORY OBJECTIVES:

I. To analyze PD-L1 expression on acute myeloid leukemia (AML) cells from peripheral blood and/or bone marrow samples at diagnosis if available and at the time of study enrollment.

II. To monitor AML minimal residual disease (MRD) by Wilms tumor 1 (WT1) polymerase chain reaction (PCR) at enrollment and at subsequent defined time points in the nivolumab-treated and control groups.

III. To perform an exploratory analysis on the frequencies, absolute numbers and subsets of T cells (including regulatory T cells) in the nivolumab-treated and control groups with an emphasis on activation markers.

IV. To perform deep sequencing of T cell receptor (TCR)-alpha and TCR-beta chains on polyclonal T cells at baseline and at subsequent time points in the nivolumab and control groups.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive nivolumab intravenously (IV) over 30 minutes once every 2 weeks. Treatment repeats every 2 weeks for 46 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo bone marrow biopsy at screening, months 3, 6, and 12, as clinically indicated, and at the time off study. Patients also undergo collection of blood samples at screening, weeks 9, 13, 25, and 53, and during off-study evaluation or at time of clinically suspected relapse. Patients may undergo echocardiography (ECHO) as clinically indicated.

ARM II: Patients undergo standard of care clinical observation for up to 2 years. Upon disease relapse, patients may cross-over to Arm I. Patients also undergo bone marrow biopsy at screening, months 3, 6, and 12, as clinically indicated, and during off-study evaluation. Patients also undergo collection of blood samples at screening, weeks 9, 13, 25, and 53, and during off-study evaluation or at time of clinically suspected relapse. Patients may undergo ECHO as clinically indicated.

After completion of study treatment, patients are followed up periodically for 2 years, every 6 months for 1 year, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

* AML patients in first complete remission (CR) (CR1) or first complete remission with incomplete blood count recovery (CRi) after induction and/or consolidation chemotherapy; except young (< 60 years) AML patients in European LeukemiaNet favorable group; (Since young AML patients in the European LeukemiaNet favorable group have excellent 2 year progression free survival [PFS] at around 64%, further maintenance therapy might not provide additional benefit; thus the current trial will exclude young favorable group AML patients), patients could receive any cycle consolidation or no consolidation per the discretion by the treating physician
* Within 60 days after bone marrow biopsy confirmed remission after the patients recover from their last course of chemotherapy, the goal to consent the eligible patient prior to the remission confirmation bone marrow biopsy at the end of the planned chemotherapy); ideally, the research samples will be collected during the bone marrow biopsy, and the patient will be enrolled to the study within 2 weeks of the bone marrow biopsy; if there is delay to enroll the patient after the bone marrow biopsy and research sample collection, it is ok not to repeat bone marrow biopsy within 4 weeks, after the last bone marrow biopsy, if there is no sign of disease relapse; a repeat bone marrow biopsy should be done if the delay of enrollment is more than 4 weeks after the last bone marrow biopsy; patients with confirmed remission within 60 days after the last bone marrow biopsy, without research samples collection, should have a repeat bone marrow biopsy conducted within two weeks prior to enrolling on the study
* Patient is not a candidate for stem cell transplant due to advanced age or co-morbidities; or the enrollee does not have donor available; or the enrollee declines stem cell transplant due to personal belief; or stem cell transplant is not standard of care based on the risk category of disease
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of nivolumab in patients < 18 years of age, children are excluded from this study, but will be eligible for future pediatric trials
* Eastern Cooperative Oncology Group (ECOG)/Karnofsky performance status of 0 or 1 (Karnofsky >= 70%)
* Life expectancy of greater than 6 months
* Leukocytes >= 1,500/mcL
* Absolute neutrophil count >= 1,000/mcL
* Platelets >= 50,000/mcL or recovery to the baseline count
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN) (except patients with Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN
* Amylase and lipase =< 1.5 x ULN without any symptoms of pancreatitis
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (CrCl) >= 50 mL/min (if using the Cockcroft-Gault formula)
* The effects of nivolumab on the developing human fetus are unknown; for this reason, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; WOCBP should use an adequate method to avoid pregnancy for 23 weeks after the last dose of investigational drug nivolumab; women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of nivolumab; women must not be breastfeeding; men who are sexually active with WOCBP must use any contraceptive method with a failure rate of less than 1% per year; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; women who are not of childbearing potential (i.e., who are postmenopausal or surgically sterile as well as azoospermic men) do not require contraception
* Women of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) or who is not postmenopausal; menopause is defined clinically as 12 months of amenorrhea in a woman over 45 in the absence of other biological or physiological causes; in addition, women under the age of 55 must have a documented serum follicle stimulating hormone (FSH) level less than 40 mIU/mL
* WOCBP receiving nivolumab will be instructed to adhere to contraception for a period of 23 weeks after the last dose of investigational product; men receiving nivolumab and who are sexually active with WOCBP will be instructed to adhere to contraception for a period of 31 weeks after the last dose of investigational product; these durations have been calculated using the upper limit of the half-life for nivolumab (25 days) and are based on the protocol requirement that WOCBP use contraception for 5 half-lives plus 30 days and men who are sexually active with WOCBP use contraception for 5 half-lives plus 90 days
* Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she (or the participating partner) should inform the treating physician immediately
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events (AEs) due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Patients should be excluded if they have had prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CTLA-4 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or immune checkpoint pathways
* Patients with known central nervous system (CNS) involvement may be excluded because of poor prognosis and concerns regarding progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events; however, if CNS disease is cleared before the treatment with nivolumab, patients could be allowed if no permanent CNS damage
* History of severe hypersensitivity reaction to any monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because nivolumab is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with nivolumab, breastfeeding should be discontinued if the mother is treated with nivolumab
* Patients with known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) might be enrolled if the viral load by PCR is undetectable with/without active treatment and absolute lymphocyte count >= 350/ul
* Patients with a positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (hepatitis C virus [HCV] antibody) indicating acute or chronic infection might be enrolled if the viral load by PCR is undetectable with/without active treatment
* Patients with active autoimmune disease or history of autoimmune disease that might recur, which may affect vital organ function or require immune suppressive treatment including systemic corticosteroids, should be excluded; these include but are not limited to patients with a history of immune related neurologic disease, multiple sclerosis, autoimmune (demyelinating) neuropathy, Guillain-Barre syndrome, myasthenia gravis; systemic autoimmune disease such as systemic lupus erythematosus (SLE), connective tissue diseases, scleroderma, inflammatory bowel disease (IBD), Crohn's, ulcerative colitis, hepatitis; and patients with a history of toxic epidermal necrolysis (TEN), Stevens-Johnson syndrome, or phospholipid syndrome should be excluded because of the risk of recurrence or exacerbation of disease; patients with vitiligo, endocrine deficiencies including thyroiditis managed with replacement hormones including physiologic corticosteroids are eligible; patients with rheumatoid arthritis and other arthropathies, Sjögren's syndrome and psoriasis controlled with topical medication and patients with positive serology, such as antinuclear antibodies (ANA), anti-thyroid antibodies should be evaluated for the presence of target organ involvement and potential need for systemic treatment but should otherwise be eligible
* Patients are permitted to enroll if they have vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger (precipitating event)
* Patients should be excluded if they have a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration; inhaled or topical steroids and adrenal replacement doses =< 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease; patients are permitted to use topical, ocular, intra-articular, intranasal, and inhalational corticosteroids (with minimal systemic absorption); physiologic replacement doses of systemic corticosteroids are permitted, even if =< 10 mg/day prednisone equivalents; a brief course of corticosteroids for prophylaxis (e.g., contrast dye allergy) or for treatment of non-autoimmune conditions (e.g., delayed-type hypersensitivity reaction caused by contact allergen) is permitted
* Patients who have had evidence of active or acute diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction and abdominal carcinomatosis which are known risk factors for bowel perforation should be evaluated for the potential need for additional treatment before coming on study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-07-02 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2026-10-08 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy Stock, Principal Investigator — University of Chicago Comprehensive Cancer Center EDDOP
Locations (46):
- United States (45):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - Smilow Cancer Center/Yale-New Haven Hospital, New Haven, Connecticut
  - Yale University, New Haven, Connecticut
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center-International Plaza, Tampa, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - University of Kansas Cancer Center, Kansas City, Kansas
  - University of Kansas Hospital-Westwood Cancer Center, Westwood, Kansas
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - NCI - Center for Cancer Research, Bethesda, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center/Dartmouth Cancer Center, Lebanon, New Hampshire
  - Rutgers Cancer Institute of New Jersey-Robert Wood Johnson University Hospital, New Brunswick, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Montefiore Medical Center-Einstein Campus, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Baylor College of Medicine/Dan L Duncan Comprehensive Cancer Center, Houston, Texas
  - Ben Taub General Hospital, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pyzer AR, Dillon LW, Sharon E, Karrison TG, Zha Y, Fulton N, Gui G, Andrew G, Streicher H, Sweet K, Yaghmour G, Liu JJ, Jonas BA, Schimmer AD, Grant S, Zeidan AM, Hildebrandt GC, Lowrey CH, Mattison RJ, Palmisiano N, Salhotra A, Tzachanis D, Baer MR, Lin TL, Patel P, Chen H, Stadler WM, Odenike O, Larson RA, Gajewski TF, Hourigan CS, Stock W, Liu H. Randomized phase 2 study to assess the role of single-agent nivolumab to maintain remission in acute myeloid leukemia. Blood Adv. 2025 May 13;9(9):2144-2152. doi: 10.1182/bloodadvances.2024015176. PMID 39928953
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Nivolumab): Patients receive nivolumab IV over 60 minutes once every 2 weeks. Treatment repeats every 2 weeks for 46 cycles in the absence of disease progression or unacceptable toxicity.
- Arm II (Observation): Patients undergo standard of care clinical observation for up to 2 years. Upon disease relapse, patients may cross-over to Arm I.
Period: Overall Study
Arm/Group | Arm I (Nivolumab) | Arm II (Observation)
Started | 41 | 41
Completed | 38 | 41
Not Completed | 3 | 0
Not completed — Protocol Violation | 2 | 0
Not completed — Never received study treatment | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Nivolumab) | Arm II (Observation) | Total
Number analyzed (Participants) | 38 | 41 | 79
Age, Continuous [Mean (Full Range); unit: years] | 63.2 [29 to 76] | 65.5 [31 to 80] | 64.4 [29 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 19 | 37
  Male | 20 | 22 | 42
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 5 | 7
  White | 32 | 32 | 64
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 4 | 6
Region of Enrollment [Number; unit: participants]
  United States | 38 | 41 | 79

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: Time from randomization to disease relapse or death from any cause
Time Frame: Assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (Nivolumab) | Arm II (Observation)
Number analyzed (Participants) | 38 | 41
months | 13.2 [8.5 to 21.8] | 10.9 [5.4 to 14.9]
Statistical Analysis 1: Comparison: Arm I (Nivolumab) vs Arm II (Observation); Test type: Superiority; p = 0.38, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.54 to 1.56]

2. Secondary Outcome: Overall Survival (OS)
Description: Time from randomization to the date of death from any cause
Time Frame: Assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm I (Nivolumab) | Arm II (Observation)
Number analyzed (Participants) | 38 | 41
Months | 53.9 [23.4 to NA] — NA = Upper confidence limit cannot be estimated due to insufficient number of participants with events | 30.9 [14.4 to NA] — NA = Upper confidence limit cannot be estimated due to insufficient number of participants with events
Statistical Analysis 1: Comparison: Arm I (Nivolumab) vs Arm II (Observation); Test type: Superiority; p = 0.23, Log Rank — One-sided p-value; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.40 to 1.51]

3. Secondary Outcome: Non-relapse Mortality (NRM)
Description: Patient death due to reasons other than relapse
Time Frame: Assessed up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab) | Arm II (Observation)
Number analyzed (Participants) | 38 | 41
Participants | 2 | 1

4. Secondary Outcome: Incidence of Adverse Effects of Nivolumab
Description: Will be assessed using National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Grade 3 or higher regardless of attribution.
Time Frame: Up to 5 years
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (Nivolumab) | Arm II (Observation)
Number analyzed (Participants) | 38 | 41
Participants | 27 | 5
Statistical Analysis 1: Comparison: Arm I (Nivolumab) vs Arm II (Observation); Test type: Superiority; p < 0.001, Fisher Exact

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Arm I (Nivolumab) | Arm II (Observation)
All-Cause Mortality (participants affected / at risk) | 16/38 | 20/41
Serious Adverse Events (participants affected / at risk) | 8/38 | 3/41
Other Adverse Events (participants affected / at risk) | 37/38 | 8/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nivolumab) (N=38) | Arm II (Observation) (N=41)
Alanine aminotransferase (ALT) increased (Investigations) | 1 | 0
Aspartate aminotransferase increase (Investigations) | 1 | 0
Confusion (Psychiatric disorders) | 1 | 0
Lung infection (Infections and infestations) | 2 | 0
Diverticulitis (Gastrointestinal disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Nivolumab) (N=38) | Arm II (Observation) (N=41)
Abdominal pain (Gastrointestinal disorders) | 5 | 1
Activated partial thromboplastin time prolonged (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 11 | 1
Alkaline phosphatase increased (Investigations) | 5 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Anemia (Blood and lymphatic system disorders) | 14 | 4
Anorexia (Metabolism and nutrition disorders) | 2 | 2
Anxiety (Psychiatric disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Aspartate aminotransferase increased (Investigations) | 13 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 0
Blood bilirubin increased (Investigations) | 2 | 2
Bruising (Injury, poisoning and procedural complications) | 4 | 1
Chills (General disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 5 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Creatinine increased (Investigations) | 5 | 1
Diarrhea (Gastrointestinal disorders) | 13 | 2
Dizziness (Nervous system disorders) | 5 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 3 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Ear pain (Ear and labyrinth disorders) | 2 | 0
Edema limbs (General disorders) | 5 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0
Fatigue (General disorders) | 16 | 3
Fever (General disorders) | 3 | 1
Flu like symptoms (General disorders) | 5 | 0
Flushing (Vascular disorders) | 3 | 0
Gastroesohpageal reflux (Gastrointestinal disorders) | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Headache (Nervous system disorders) | 8 | 1
Hematuria (Renal and urinary disorders) | 2 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 2 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 12 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3 | 1
Hypertension (Vascular disorders) | 14 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 2 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 2
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatremia (Metabolism and nutrition disorders) | 3 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 7 | 3
Hypothyroidism (Endocrine disorders) | 7 | 0
Infusion related reaction (General disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 3 | 2
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lipase increased (Investigations) | 5 | 0
Lymphocyte count decreased (Investigations) | 8 | 5
Mucositis oral (Gastrointestinal disorders) | 4 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Nausea (Gastrointestinal disorders) | 11 | 0
Neutrophil count decreased (Investigations) | 12 | 4
Pain (General disorders) | 5 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Paresthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 3 | 2
Platelet count decreased (Investigations) | 14 | 7
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 7 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 9 | 2
Serum amylase increased (Investigations) | 4 | 0
Toothache (Gastrointestinal disorders) | 2 | 0
Upper respiratory infection (Infections and infestations) | 2 | 0
Vomiting (Gastrointestinal disorders) | 5 | 0
Weight gain (Investigations) | 5 | 0
White blood cell decreased (Investigations) | 12 | 7
Shoulder pain (Musculoskeletal and connective tissue disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02275533/Prot_SAP_000.pdf
  • Informed Consent Form (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/33/NCT02275533/ICF_001.pdf